CLINICAL TRIAL: NCT02918240
Title: The Effect of Different Appointment Intervals on Treatment Time in Patients Receiving Orthodontic Treatment With Fixed Appliances
Brief Title: How Often Should We See Our Orthodontic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/LO/0522
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2020-09

CONDITIONS: Orthodontics

ARMS (4):
- 4 week interval (Experimental): Patients will be seen every 4 weeks to adjust their orthodontic braces
  Interventions: Procedure: Appointment intervals; Device: fixed orthodontic braces
- 6 week interval (Experimental): Patients will be seen every 6 weeks to adjust their orthodontic braces
  Interventions: Procedure: Appointment intervals; Device: fixed orthodontic braces
- 8 week interval (Experimental): Patients will be seen every 8 weeks to adjust their orthodontic braces
  Interventions: Procedure: Appointment intervals; Device: fixed orthodontic braces
- 10 week interval (Experimental): Patients will be seen every 10 weeks to adjust their orthodontic braces
  Interventions: Procedure: Appointment intervals; Device: fixed orthodontic braces

INTERVENTIONS:
Procedure: Appointment intervals
Device: fixed orthodontic braces

SUMMARY:
Fixed orthodontic braces are routinely used to straighten teeth and correct the bite of individuals. Once the braces are fit, the patient is recalled every few weeks to adjust or tighten the brace. Although convention states that the patient returns every 6-8 weeks to have the brace adjusted, there is no consensus or evidence to support a specific timeframe. Indeed some orthodontist see their patients as frequently as every 4 weeks and others as long as every 10 weeks. The aim of this investigation is to determine whether the amount of time between brace adjustment appointments has an effect on the overall treatment time. Knowing which appointment interval will lead to the shortest overall treatment time will be of benefit to patients as prolonged orthodontic treatment may be associated with an increased incidence of adverse effects associated with orthodontic treatment.

Patients who are to be treated with fixed orthodontic braces at will be invited to take part in the study. Consenting subjects will be randomly allocated into one of four groups. The first will be seen to adjust their brace every 4 weeks, the second group every 6 weeks, the third group every 8 weeks and the fourth group every 10 weeks.

The primary outcome measure is the total treatment time. The mean treatment time of each of the four groups will be compared to establish whether or not treatment appointment intervals affects treatment time.

Secondary outcome measures will include difference in number of appointments required throughout the course of treatment between groups, differences in treatment outcomes, differences in patient compliance.

DETAILED DESCRIPTION:
Patients at Grosvenor House Orthodontic Practice who are to be treated with fixed orthodontic appliances and fulfil the inclusion criteria will be invited to participate in the research.

Once consented, patients will be randomly allocated to one of four groups, each group specifying a different amount of time between appointments following brace fitting.

Once the subject has had their fixed orthodontic appliance fit, they will be offered appointments every 4 weeks, 6 weeks, 8 weeks or 10 weeks to adjust there brace, depending on which group they are in.

All patients will have both arches bonded simultaneously in a standardized way using 3M Unitek pre-coated Gemini brackets with MBT prescription. The initial archwire will be 0.014 nickel titanium ligated using standard elastomeric ligation. Patients will then progress to 0.018 nickel titanium followed by 0.019x0.025 heat activated nickel titanium followed by 0.019x0.025 stainless steel. Round stainless steel archwires will be permitted if indicated for finishing or as a lower working archwire in Class III patients but the original archwire sequence will be adhered to wherever possible. Progression to the next archwire will only occur once each archwire becomes passive.

Space closure of extraction spaces where indicated will be done with E-Links (TP Orthodontics, Inc.) running from the hook on the molar tube to a hook crimped onto the archwire between the lateral incisor and canine.

Patients who fail to attend or cancel appointments will be offered another appointment within 1 week of the original appointment.

Once the orthodontic treatment is complete to the satisfaction of the patient and orthodontist, the brace will be removed. The time in days from brace fit to brace removal will be noted and a total treatment time will be recorded for each subject. A comparison will be made on the total treatment time between the four groups.

A basic oral hygiene examination will be done at each appointment. The data will be analysed following treatment to determine whether appointment frequency has an impact on oral hygiene.

A record will also be made of the number of appointments missed or cancelled and a comparison between groups will be made during the analysis.

Treatment outcomes will be determined using the PAR (peer assessment rating) system which assesses certain features of the occlusion from pre treatment and post treatment plaster models, quantifying the level of improvement brought about by treatment. The outcome of treatment, as measured by PAR, will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Children who are to be treated with upper and lower fixed orthodontic appliances
2. Aged between 10 and 18 years old at start of treatment
3. Consent to participating in trial

Exclusion Criteria:

* Patients requiring functional orthodontic appliances
* Presence of unerupted impacted teeth
* Presence of deciduous teeth
* Hypodontia excluding absent third molars
* Any craniofacial anomalies
* Medical contraindications

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Total Treatment Time | 2 years
  Time between fitting braces and removing braces

SECONDARY OUTCOMES:
Number of appointments needed | 2 years
  Total clinical time used
Patient compliance survey | 2 years
  This will be measured by comparing oral hygiene, failed/cancelled appointment and broken braces between groups
Treatment Outcome | 2 years
  PAR scores will be used to compare outcome between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Grosvenor House Orthodontic Practice, Royal Tunbridge Wells, Kent, United Kingdom